CLINICAL TRIAL: NCT00076453
Title: Clinical Effects of Altered Biomechanics in Knee Osteoarthritis
Brief Title: A Study of Orthotic Shoe Inserts for Controlling Osteoarthritic Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Joel A. Block, MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIAMS-116; 2P50AR039239-16 (NIH)
Record Dates: First submitted 2004-01-22; First posted 2004-01-26 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Osteoarthritis
Keywords: Knee Pain; Degenerative Arthritis; Cartilage Disease; Non-drug Therapy
MeSH Terms: conditions — Osteoarthritis; Cartilage Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will wear lateral wedge orthotic inserts.
  Interventions: Device: Lateral wedge orthotic shoe inserts
- 2 (Active Comparator): Participants will wear standard orthotic inserts.
  Interventions: Device: Standard orthotic shoe inserts

INTERVENTIONS:
Device: Lateral wedge orthotic shoe inserts — Customized lateral wedge orthotic shoe inserts
  Arms: 1
Device: Standard orthotic shoe inserts — Neutral orthotic inserts
  Arms: 2

SUMMARY:
Osteoarthritis is a degenerative joint disease and is the most common form of arthritis. This study will evaluate the effectiveness of customized shoe inserts in controlling and relieving the pain of knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a chronic disease causing deterioration of the joint cartilage and the formation of bone spurs at the margins of the joints. Knee OA causes substantial pain, suffering, and disability, as well as enormous economic burden on the patient; unfortunately, treatment provides relief but not a cure. The majority of patients with symptomatic knee OA do not attain satisfactory long-term relief, even with recent advances in pain relievers. Analgesic treatment may relieve the pain but does not improve biomechanics and may even aggravate OA.

Although OA is complex and not completely understood, disease onset and progression are at least partly related to responses by bone and cartilage to biomechanical loading. Devices that promote pressure reduction from the medial knee may provide pain relief while simultaneously protecting the joint from further degeneration; one such device is a lateral wedge orthotic shoe insert. When worn during weight-bearing activity, these inserts have been shown to reduce loading of the medial compartment and may provide pain relief. This study will evaluate the effectiveness of orthotic shoe inserts in controlling and relieving knee OA. The study will also assess improvements in loading biomechanics of the knee.

This is a 3-year study. Patients will be randomly assigned to one of two groups; the first group will receive lateral wedge orthotic inserts and the second group will receive standard orthotic inserts. There will be 10 study visits during the course of the study. Patients will undergo X-rays and bone mineral density testing (DEXA) and 3 blood collections during the course of the study.

ELIGIBILITY:
Inclusion Criteria

* Able and willing to give informed consent and to comply with the study protocol and follow-up instructions
* Symptomatic and radiographic OA of the knee
* Knee pain upon walking
* Predominant medial compartment OA

Exclusion Criteria

* Knee flexion contracture of greater than 15 degrees or inability to walk without assistance
* Predominant lateral compartment OA of either knee
* Greater than 3 degree valgus or greater than 12 degree varus deformity of either knee, as defined by the mechanical axis
* Clinically evident OA of the ankle or hip
* Clinically significant intrinsic foot disease upon podiatric evaluation, including any foot condition that may be aggravated by wearing orthotics
* Substantial obesity, defined as having body mass index (BMI) greater than 35
* Anticipation of surgery involving any joint of either lower extremity in the next 3 years
* Habitual use of inappropriate shoewear that would interfere with adequate use of the orthotic inserts
* Inflammatory arthropathy, such as rheumatoid arthritis, systemic lupus, or active gout
* Chronic infection in any joint of the lower extremities
* History of fracture of either lower extremity within 6 months of study entry
* History of knee or hip arthroplasty or of surgical arthroscopy of either knee within 3 months of study entry
* History of intra-articular injections (glucocorticoids or hyaluronic acid derivatives) in the index knee within 6 months of study entry
* Pregnancy
* Any medical condition which, in the opinion of the investigator, would render the patient unable to comply with the protocol

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Pain reduction | Years 2 and 3

SECONDARY OUTCOMES:
Reduction in loading of the medial knee | Years 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Joel A. Block, MD, Principal Investigator — Rush University Medical Center, Section of Rheumatology
Locations (1):
- Rush University Medical Center, Section of Rheumatology, Chicago, Illinois, United States

REFERENCES:
- [Derived] Tezcan ME, Goker B, Lidtke R, Block JA. Long-term effects of lateral wedge orthotics on hip and ankle joint space widths. Gait Posture. 2017 Jan;51:36-40. doi: 10.1016/j.gaitpost.2016.09.017. Epub 2016 Sep 21. PMID 27693959